CLINICAL TRIAL: NCT05768698
Title: Valutazione Delle Pressioni di Riempimento Del Ventricolo Sinistro Attraverso l'Impiego di un Software di Intelligenza Artificiale Applicato Alla Stima Dello Strain Atriale Sinistro Con Ecocardiografia Speckletracking: Studio di Validazione Mediante Cateterismo Cardiaco
Brief Title: Assessment of Left Ventricular Filling Pressure by Applying Artificial Intelligence Algorithms to Left Atrial Speckle-tracking Echocardiography
Acronym: LVEDP
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 09V102
Record Dates: First submitted 2023-02-22; First posted 2023-03-14 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure, Diastolic; Echocardiography
Keywords: Transthoracic echocardiography; left ventricular filling pressure; artificial intelligence; right heart catheterization
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Software algorithm — Validation of a software package based on an artificial intelligence algorithm for automated non-invasive estimation of LVFP against invasively measured ones by left and right heart catheterization

SUMMARY:
The goal of this single-center, prospective, observational study is to validate a software package based on an artificial intelligence algorithm for automated non-invasive estimation of LVFP against invasively measured ones by left and right heart catheterization; In addition, the added value of this new automated software to detect increased LVEDP > 15 mm Hg compared to the current ASE/EACVI algorithm for assessing diastolic dysfunction and longitudinal left atrial strain during the reservoir phase will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 yo,
* Signed informed consent to be part of this study,
* No pregnancy,
* Good acoustic window and patient cooperation to obtain good 2- and 3-dimensional datasets focused on left atrium (LA),

Exclusion Criteria:

* Unwillingness to be part of the study,
* Patients with poor 2-dimensional imaging quality in ≥ 1 LA segment or lacking of a discernible R-R interval, which might preclude accurate strain measurements,
* Patients with more than mild mitral valve heart disease, aortic regurgitation, left side valvular prosthesis or mitral valve repair, mitral annulus calcification (≥ 5 mm),
* Patients with history or presence of atrial fibrillation (AF), supraventricular arrhythmias, ventricular paced rhythm, left bundle branch block (LBBB),
* Patients taking diuretics or vasodilators (nitrates) on the day of the examination, which could alter loading conditions.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred to our cath lab for clinically indicated coronary angiography or right heart catheterization for the diagnosis of dyspnea
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2024-06-11 (Estimated); Study Completion 2024-06-11 (Estimated)

PRIMARY OUTCOMES:
Left ventricular filling pressure | During procedure
  Invasively measured left ventricular filling pressure by right heart catheterization

CONTACTS AND LOCATIONS:
Locations (1):
- Philips Healthcare, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Available only upon reasonable request to study P.I.